CLINICAL TRIAL: NCT05435794
Title: Long-term Benefits of Continuous Positive Pressure Therapy or Mandibular Advancement Devise on the Sleep of Patients With Obstructive Sleep Apnea
Brief Title: Long-term Benefits of CPAP or MAD Treatment on the Sleep of OSAS Patients
Acronym: REMAP
Status: Recruiting | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00629-34
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: OSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient treated with CPAP
  Interventions: Device: CPAP
- Patient treated with MAD
  Interventions: Device: MAD

INTERVENTIONS:
Device: CPAP — Fixed-pressure CPAP device for the treatment of sleep apnea with optional humidification and heated circuit. This device is a Class II device. It has a remote monitoring function allowing service providers to track the use of the device.
  Groups: Patient treated with CPAP
Device: MAD — mandibular device orthosis made to measure from the dental impressions of patients, made by the specialist in the masticatory apparatus for the treatment of sleep apnea.
  Groups: Patient treated with MAD

SUMMARY:
The REMAP study aims to follow a cohort of 400 patients in around ten sleep centers in France and to collect clinical routine data. The objectives of this study are to investigate the effects of one-year management of OSA by CPAP or MAD on sleep architecture defined by objective macro and micro sleep architecture parameters using a sleep test device. sleep connected at home, to assess the quality of sleep and the quality of life reported by patients. The study will also allow us to define predictive factors for improving sleep quality during OSA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient already included in the SunSAS study (No. ID/RCB: 2021-A01827-34) or Patient who has undergone polygraphy or polysomnography eligible for treatment with CPAP or MAD in the context of OSA.
* Patient with a sleep test performed with the Sunrise device
* Men or Women from 18 to 80 years old
* Patient with OSAS eligible for CPAP or MAD therapy
* Affiliated patient or beneficiary of a social security scheme
* Signed informed consent

Exclusion Criteria:

* Patient previously treated for OSAS by CPAP or MAD during the last five years
* Patient with COPD or other respiratory diseases.
* Patient with contraindications to PPC or MAD therapy
* Patient with unstable heart disease or New York Heart Association class III or IV heart failure
* Patient unable to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited based on scheduled appointments at the various centers that participate in the SunSAS clinical trial and are diagnosed and managed for their OSA in accordance with standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
To determine the evolution of deep slow-wave sleep at one year in OSA patients according to the treatment initiated by continuous positive pressure or mandibular advancement device (MAD). | 12 months
  Objective evolution of deep slow-wave sleep time. Changes collected with a home-connected sleep testing device by comparing data from the initial visit (diagnosis) with data collected at 12 months (± 2 weeks) in a patient treated with CPAP or MAD.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - CHU Lyon - Hôpital de la Croix-Rousse, Lyon
  - Hopital Europeen Marseille, Marseille
  - APHP - Pitié-Salpêtrière University Hospital, Paris
  - AP-HP Bichat, Paris
  - CHU Reims, Reims
  - Polyclinique St Laurent, Rennes
  - Centre du Sommeil, Saint-Martin-d'Hères